CLINICAL TRIAL: NCT01607814
Title: Oxidative Stress and Haemostasis Abnormalities in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Director, Head of Internal Medicine, Principal Investigator, Clinical Professor, University of Roma La Sapienza
Other Study IDs: Cirrhosis and Oxidative Stress
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Cirrhosis
Keywords: cirrhosis; oxidative stress; NADPH oxidase; isoprostanes; PUFA balance; platelet activation; coagulation abnormalities
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum and urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cirrhotic Patients: Patients affected by cirrhosis of any etiology and severity
- Control Group: Subjects age, sex and comorbidities matched

SUMMARY:
Patients with cirrhosis can have abnormalities in laboratory tests reflecting changes in primary and secondary haemostasis.

Such changes have been considered particularly relevant in the bleeding complications that occur in cirrhosis.

However, several studies have shown that routine diagnostic tests are not clinically useful to stratify bleeding risk in patients with cirrhosis. Moreover, treatments used to increase platelet count or to modulate platelet function could potentially do harm. Consequently the optimal management of bleeding complications is still a matter of discussion.

Moreover, in the last two decades there has been an increased recognition that not only bleeding but also thrombosis complicates the clinical course of cirrhosis. Over the last years, emerge that in vivo platelet function and coagulation cascade might be modulated by an alteration of pro-oxidant and antioxidant balance. Thus It has previously been demonstrated that chronic liver diseases are characterized by increased oxidative stress state.

Aim of the study is to analyse the relationship between oxidative stress, haemostatic balance and clinical complications in cirrhosis.

DETAILED DESCRIPTION:
Natural history of cirrhotic patients is complicated by gastrointestinal bleeding which remains the most dramatic event considering is acute onset and is negative impact on life expectancy of LC patient. Over the last decade, improvements in therapy produce a sensible reduction in mortality of at least 20% at 6 weeks (8% at 24 hours) for each one episode of gastrointestinal bleeding.

Furthermore, portal vein thrombosis (PVT) is a frequent (10-20%) event in liver cirrhosis (LC), often asymptomatic, which may worsen its clinical course by favouring gastrointestinal bleeding, in particular precipitating the grade of portal hypertension.

Standing the coexistence of thrombotic and bleeding manifestations of difficult interpretation and management, only the elucidation of the mechanism leading to this complex hemostatic disturbance occurring in LC, would help us to explore new therapeutic strategies to prevent bleeding improving clinical outcomes.

However the mechanisms underlying specific cirrhotic hemostatic disturbance is still unclear.

On the last decade, has been investigated the presence of abnormalities in all hemostatic phases such as primary haemostasis (altered platelet function) or fibrinolysis and coagulation (impaired synthesis and activity of coagulation factors or hyperfibrinolysis.). The derangement of coagulation balance has been investigated and several studies identified abnormal haemostasis tests or coagulation factors as useful prognostic indexes of survival in LC patients Observational studies have shown that Factor VII, vitamin k dependent with short half-life (2 hours) is useful prognostic index of both acute and chronic liver insufficiency.

Less well studied and more interesting is the potential role of primary haemostasis in determination of typical thrombotic and bleeding complications..

It is well known that chronic liver disease is characterized by variable thrombocytopenia and thrombocytopathy Observational studies pointed out that platelet dysfunction is an abnormality occurring prevalently in severe liver failure. Child-Pugh C class patients present lower platelet counts and more prolonged bleeding times. Since platelets abnormalities are much more frequent depending on liver insufficiency severity, it is probably that several mechanisms account for that complex platelet dysfunction. A retrospective study with a 3 years follow- up demonstrate a strong association between previous gastrointestinal hemorrhage, prolonged bleeding time(> 10 minutes) and lower platelet count (<100.000/ μl) without explaining if this relationship is a casual one. These data indicate that in LC patients with an history of gastrointestinal blood loss thrombocytopenia or/and thrombocytopathy might be determinant in acute phase of bleeding. However, at the moment, studies in LC patients that prospectively analyze the platelet function role in favoring hemorrhage activity are not still available.

Several hypothesis has been proposed to explain mechanisms leading to platelet abnormal function in LC patients, however, their nature and clinical significance are still a matter of discussion. For example, it is on debate whether platelet activity is influenced in positively or negatively manner in LC patients.

From literature emerges that there is no agreement on the mechanism leading in-vivo platelet aggregation in patients affected by chronic liver disease. Laffi et al. suggested that in cirrhotic patients defective aggregation is most likely dependent on the alteration of the transmembrane signaling pathways and the increased urinary excretion of systemic TXA2 metabolites may be related to increased intrasplenic platelet destruction. On the contrary , Davì et al. found a significant correlation between urinary excretion of 2,3-dinor thromboxane B2(TXB2) and plasma prothrombin fragment 1+2 (F1+2), suggesting that clotting activation could partly account for in vivo platelet activation.

Moreover, increased soluble P-selectin levels, in vivo marker of platelets activation, were found in patients with chronic C hepatitis and were correlated with severity of disease. These findings support the hypothesis that thrombocytopenia is not only related to autoimmunity mechanism but also to a condition of in vivo platelet activation induced directly by HCV infection.

Over the last years, emerge that in vivo platelet function might be modulated by an alteration of pro-oxidant and antioxidant balance. F(2)-isoprostanes are prostaglandin F2-like compounds produced in vivo by nonenzymatic free radical-induced peroxidation of arachidonic acid in a COX-independent manner.

Unlike lipid hydroperoxides, F2-IsoPs are also specific products of free radical-induced lipid peroxidation, chemically stable compounds and detectable in plasma and urine. One of the F2-IsoPs, which have shown interestingly to induce platelet aggregation and to stimulate vascular smooth muscle cell proliferation.

The 8-iso-prostaglandin F2a measurement represent a sensible and specific index of lipid peroxidation.

It has previously been demonstrated that chronic liver diseases are characterized by increased ROS production as well as decreased activity of antioxidant systems, resulting in oxidative stress.

Hepatic fibrosis represents a wound healing response to injury that ultimately leads to cirrhosis. Mechanisms involved are still on investigation. Experimental and human studies showed that markers of oxidative stress and proinflammatory cytokines, are increased in liver diseases suggesting that inflammation could have a pivotal role in terms of progression of chronic damage.

NADPH oxidase complex has been recognized as a critical mediator of liver fibrosis while is unexplored his probably role in modulating platelet function in cirrhotic setting.

To investigate relationship between platelets, coagulation parameters and oxidative stress in cirrhotic patients, the investigators planned a cross-sectional study finalized to clarify platelets, haemostatic balance and oxidative stress contribution to thrombotic and bleeding complications occurring in cirrhosis's natural history, such as to identify new haemostatic parameters with predictive value on cirrhotic evolution and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any etiology and severity
* Signed Written Informed Consent

Exclusion Criteria:

* Treatment with non steroidal anti-inflammatory drugs or antithrombotic drugs (antiplatelets and anticoagulants)
* Vitamin Supplementation
* Pregnancy
* Cholestatic liver disease
* Hepatocarcinoma and Extrahepatic neoplasm
* Active infective or inflammatory diseases
* Recent major or minor surgery (< 3 months)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by cirrhosis of any etiology and severity
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress markers | 2 years
  Evaluate the F2-Isoprostanes, in vivo oxidative stress markers, production in cirrhotic patients and its influence on haemostatic balance.

SECONDARY OUTCOMES:
Thrombotic Events | 2 years
  Occurrence of thrombotic complications
Bleeding Events | 2 years
  Occurrence of bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — Divisione di Prima Clinica Medica - Sapienza University of Rome
Locations (1):
- Internal and Medical Specialties Department, Policlinico Umberto I, Rome, Rome, Italy